CLINICAL TRIAL: NCT01243151
Title: A Phase 1, Placebo-controlled, Randomized Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Following Multiple Intravenous Doses Of Pf-04950615 In Healthy Adult Subjects With Hypercholesterolemia
Brief Title: Safety And Tolerability Of Multiple Doses Of PF-04950615 (RN316) In Subjects With Hypercholesterolemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1481009
Record Dates: First submitted 2010-11-03; First posted 2010-11-18 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Hypercholesterolemia; Dyslipidemia
Keywords: Hypercholesterolemia; Dyslipidemia; LDL; High Cholesterol; Japanese Volunteers; PF-04950615; RN316
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Placebo Comparator)
  Interventions: Biological: PF-04950615 (RN316)
- B (Experimental)
  Interventions: Biological: PF-04950615 (RN316)
- C (Experimental)
  Interventions: Biological: PF-04950615 (RN316)
- D (Experimental)
  Interventions: Biological: PF-04950615 (RN316)
- E (Experimental)
  Interventions: Biological: PF-04950615 (RN316)

INTERVENTIONS:
Biological: PF-04950615 (RN316) — Infusion every week
  Arms: A
Biological: PF-04950615 (RN316) — Infusion every week
  Arms: B
Biological: PF-04950615 (RN316) — Infusion every week
  Arms: C
Biological: PF-04950615 (RN316) — Infusion every week
  Arms: D
Biological: PF-04950615 (RN316) — Infusion every week
  Arms: E

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of repeated doses of PF-04950615 (RN316) in study volunteers with hypercholesterolemia. PF-04950615 is an investigational drug that is currently being studied as a lipid lowering agent.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C must be greater or equal to 130 mg/dl
* BMI must be between 18.5 and 40 kg/m2
* Japanese volunteers must have 4 Japanese grand parents born in Japan

Exclusion Criteria:

* History of cardiovascular or cerebrovascular event during the past year.
* Poorly controlled type 1 or type 2 diabetes mellitus
* Subjects who have taken lipid lowering therapies within the last 3 months of screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - California Clinical Trials Medical Group, Culver City, California
  - Glendale Adventist Medical Center, Glendale, California
  - SeaView Research, Inc., Miami, Florida
  - Covance Clinical Research Unit, Inc., Honolulu, Hawaii
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Prism Research, Saint Paul, Minnesota
  - Healthcare Discoveries, LLC dba ICON Development Solutions, San Antonio, Texas

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Wan H, Gumbiner B, Joh T, Riel T, Udata C, Forgues P, Garzone PD. Effects of Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Inhibition with Bococizumab on Lipoprotein Particles in Hypercholesterolemic Subjects. Clin Ther. 2017 Nov;39(11):2243-2259.e5. doi: 10.1016/j.clinthera.2017.09.009. Epub 2017 Oct 14. PMID 29037448
- [Derived] Udata C, Garzone PD, Gumbiner B, Joh T, Liang H, Liao KH, Williams JH, Meng X. A Mechanism-Based Pharmacokinetic/Pharmacodynamic Model for Bococizumab, a Humanized Monoclonal Antibody Against Proprotein Convertase Subtilisin/Kexin Type 9, and Its Application in Early Clinical Development. J Clin Pharmacol. 2017 Jul;57(7):855-864. doi: 10.1002/jcph.867. Epub 2017 Feb 9. PMID 28181260
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481009&StudyName=Safety%20And%20Tolerability%20Of%20Multiple%20Doses%20Of%20PF-04950615%20%28RN316%29%20In%20Subjects%20With%20Hypercholesterolemia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to PF-04950615 once daily on Day 1, 8, 15 and 22 in 28 days treatment period.
- PF-04950615 0.25 mg/kg: Participants received PF-04950615 0.25 milligram per kilogram (mg/kg), intravenous (IV) infusion once daily on Day 1, 8, 15 and 22 in 28 days treatment period.
- PF-04950615 0.50 mg/kg: Participants received PF-04950615 0.50 mg/kg, IV infusion once daily on Day 1, 8, 15 and 22 in 28 days treatment period.
- PF-04950615 1.0 mg/kg: Participants received PF-04950615 1.0 mg/kg, IV infusion once daily on Day 1, 8, 15 and 22 in 28 days treatment period.
- PF-04950615 1.5 mg/kg: Participants received PF-04950615 1.5 mg/kg, IV infusion once daily on Day 1, 8, 15 and 22 in 28 days treatment period.
Period: Overall Study
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.5 mg/kg
Started | 12 | 14 | 14 | 14 | 14
Treated | 12 | 14 | 14 | 13 | 14
Completed | 12 | 13 | 13 | 12 | 14
Not Completed | 0 | 1 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0
Not completed — Randomized but not treated | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- PF-04950615 1.50 mg/kg: Participants received a single dose of PF-04950615 1.50 milligram/kilogram (mg/kg), intravenous (IV) infusion once on Day 1,8,15 and 22.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg | Total
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (13.7) | 52.0 (7.8) | 51.5 (13.0) | 52.5 (14.3) | 55.1 (8.8) | 53.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 4 | 5 | 6 | 27
  Male | 6 | 8 | 10 | 8 | 8 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting and Intolerable Treatment-Related Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Dose limiting and intolerable treatment-related AEs were the AEs resulting from drug overdose, drug withdrawal, drug abuse, drug misuse, drug interactions, drug dependency, extravasation, exposure in utero, exposure during breast feeding.
Time Frame: Baseline up to Follow-up period (Day 78)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
participants
  With dose limiting treatment related AEs | 0 | 0 | 0 | 0 | 0
  With intolerable treatment related AEs | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Treatment-Related Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to Day 78 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Follow-up period (Day 78)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
participants
  Treatment emergent AEs | 9 | 8 | 5 | 7 | 9
  Treatment emergent SAEs | 0 | 1 | 0 | 0 | 0
  Treatment related AEs | 3 | 6 | 3 | 2 | 5

3. Primary Outcome: Number of Participants With Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug. AE was assessed according to common terminology criteria for adverse events (CTCAE) version 4.0 severity grades- Grade 1: mild (asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated); Grade 2: moderate (minimal, local or non invasive intervention indicated); Grade 3: severe (medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling); Grade 4: Life-threatening consequences; urgent intervention indicated and Grade 5: Death related to AE.
Time Frame: Baseline up to Follow-up period (Day 78)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
participants
  Grade 1 | 8 | 7 | 5 | 5 | 6
  Grade 2 | 1 | 0 | 0 | 2 | 3
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 2 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria: Haemoglobin(Hgb), hematocrit, RBC: <0.8*lower limit of normal(LLN),mean corpuscular volume, mean corpuscular Hgb concentration <0.9*LLN or>1.1*upper limit of normal(ULN), platelet<0.5*LLN or>1.75*ULN, WBC<0.6*LLN or>1.5*ULN, lymphocyte, neutrophil<0.8*LLN or>1.2*ULN, basophil, eosinophil, monocyte>1.2*ULN; bilirubin>1.5*ULN, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma glutamyl transferase, lactate dehydrogenase>3.0*ULN,total protein,albumin<0.8*LLN or>1.2*ULN; blood urea nitrogen, creatinine>1.3*ULN,uric acid>1.2*ULN;sodium<0.95*LLNor>1.05*ULN,potassium,chloride,calcium,bicarbonate<0.9*LLN or>1.1*ULN; glucose<0.6*LLN or >1.5*ULN, urine specific gravity<1.003 or>1.030,urine pH<4.5or>8,urine glucose, ketones, urine protein,urine blood/Hgb,urobilinogen,bilirubin,nitrite, leukocyte esterase>=1; urine RBC,WBC>=20,urine epithelial cells>=6,urine granular casts,hyaline casts>1,urine bacteria>20,partial thromboplastin time,prothrombin:>1.1*ULN.
Time Frame: Baseline up to Follow-up period (Day 78)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
participants | 7 | 10 | 2 | 7 | 7

5. Primary Outcome: Number of Participants With Clinically Relevant Changes in Vital Signs
Description: Criteria for clinically relevant vital signs: supine and standing systolic blood pressure (SBP): less than (<) 90 millimeter of mercury (mmHg); supine and standing diastolic blood pressure (DBP): <50 mmHg. Maximum increase from baseline (IFB) or decrease from baseline (DFB) in supine and standing SBP: greater than or equal to (>=) 30 mmHg and maximum IFB or DFB in supine and standing DBP: >=20 mmHg. Supine pulse rate: <40 and greater than (>) 120 beats per minute (bpm); standing pulse rate: <40 and >140 bpm.
Time Frame: Baseline up to Follow-up period (Day 78)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
participants
  Supine SBP | 1 | 0 | 0 | 0 | 0
  Maximum IFB in standing SBP | 4 | 2 | 1 | 1 | 2
  Maximum IFB in supine DBP | 2 | 0 | 2 | 0 | 1
  Maximum IFB in standing DBP | 1 | 1 | 0 | 1 | 1
  Maximum DFB in supine SBP | 1 | 1 | 1 | 1 | 1
  Maximum DFB in standing SBP | 0 | 2 | 4 | 0 | 0
  Maximum DFB in supine DBP | 0 | 1 | 1 | 1 | 1
  Maximum DFB in standing DBP | 2 | 2 | 3 | 4 | 0
  Standing SBP | 1 | 1 | 0 | 0 | 3
  Supine DBP | 0 | 0 | 0 | 0 | 0
  Standing DBP | 0 | 0 | 0 | 0 | 0
  Supine Pulse Rate | 0 | 0 | 0 | 0 | 0
  Standing Pulse Rate | 0 | 0 | 0 | 0 | 0
  Maximum IFB in supine SBP | 2 | 0 | 2 | 2 | 2

6. Primary Outcome: Number of Participants With Clinically Relevant Changes in Electrocardiogram (ECG) Parameters
Description: Criteria for clinically relevant ECG parameters: PR interval: maximum IFB of >=25 percent or 50 percent; QRS complex: maximum IFB of >=25 or 50 percent; QTcF interval (Fridericia's Correction): maximum IFB of >=30 millisecond (msec) to <60 msec and maximum IFB of >=60 msec.
Time Frame: Baseline up to Follow-up period (Day 78)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
participants
  PR interval: Maximum IFB | 1 | 0 | 0 | 0 | 0
  QRS Complex: Maximum IFB | 0 | 0 | 0 | 0 | 0
  QTcF Interval: Maximum IFB >=30 to <60 msec | 0 | 2 | 0 | 1 | 2
  QTcF Interval: Maximum IFB >=60 msec | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Anti-drug Antibodies (ADA)
Description: The number of participants with at least one positive ADA were summarized for each treatment arm. Participants with positive antibody titer of >4.32 milligram/milliliter (mg/mL) were considered as ADA positive.
Time Frame: Baseline up to Follow-up period (Day 78)
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Only the participants who received a dose of PF-04950615 0.25, 0.50, 1.0, and 1.50 mg/kg were planned to be analysed for this outcome measure.
Measure: Number; unit: participants
Arm/Group | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 14 | 14 | 13 | 14
participants | 0 | 1 | 1 | 2

8. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-04950615
Description: AUCtau is area under the concentration-time profile from time zero to time tau (τ), the dosing interval, where tau =168 hours.
Time Frame: Day 1 and 22: pre-dose and 1, 6, 9, 24 and 72 hours post dose
Population: Pharmacokinetic (PK) parameter analysis population included all enrolled participants who were treated and had at least 1 of the PK parameters of interest. Here 'n' signifies those participants who were evaluable at the specified time points for each reporting group, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/ milliliter (ng*h/mL)
Arm/Group | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 14 | 14 | 13 | 14
nanogram*hour/ milliliter (ng*h/mL)
  Day 1 | 596700 (13) | 1224000 (23) | 2697000 (14) | 4253000 (18)
  Day 22: number analyzed (Participants) | 13 | 13 | 12 | 14
  Day 22 | 749800 (12) | 2134000 (22) | 4766000 (26) | 8351000 (16)

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04950615
Description: Tmax is the time at which maximum plasma concentration (Cmax) occurred.
Time Frame: Day 1 and 22: pre-dose and 1, 6, 9, 24 and 72 hours post dose
Population: PK parameter analysis population included all enrolled participants who were treated and had at least 1 of the PK parameters of interest. Here 'n' signifies those participants who were evaluable at the specified time points for each reporting group, respectively.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 14 | 14 | 13 | 14
hour
  Day 1 | 6.00 [0.883 to 9.00] | 3.61 [1.00 to 24.00] | 1.00 [0.867 to 9.18] | 1.00 [0.833 to 24.00]
  Day 22: number analyzed (Participants) | 13 | 13 | 12 | 14
  Day 22 | 6.00 [0.850 to 9.00] | 1.30 [0.867 to 9.00] | 6.00 [0.850 to 24.00] | 6.00 [0.850 to 9.00]

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04950615
Time Frame: Day 1 and 22: pre-dose and 1, 6, 9, 24 and 72 hours post dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 14 | 14 | 13 | 14
nanogram per milliliter (ng/mL)
  Day 1 | 8077 (19) | 15080 (20) | 31380 (13) | 45110 (15)
  Day 22: number analyzed (Participants) | 13 | 13 | 12 | 14
  Day 22 | 10170 (11) | 23680 (50) | 45820 (17) | 76180 (15)

11. Secondary Outcome: Plasma Decay Half-Life (t1/2) of PF-04950615
Description: t1/2 was the time measured for the plasma concentration of PF-04950615 to decrease by one half. t1/2 was calculated as Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Day 1 and 22: pre-dose and 1, 6, 9, 24 and 72 hours post dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 14 | 14 | 13 | 14
hour
  Day 1: number analyzed (Participants) | 13 | 0 | 1 | 0
  Day 1 | 50.39 (6.4231) |  | 71.50 (NA) — Standard deviation was not calculated as only 1 participant was evaluable. |
  Day 22: number analyzed (Participants) | 11 | 13 | 11 | 13
  Day 22 | 94.24 (57.042) | 140.4 (45.610) | 155.6 (38.503) | 247.2 (85.361)

12. Secondary Outcome: Apparent Clearance (CL) of PF-04950615
Description: CL was calculated as Dose/AUCtau. AUCtau is area under the concentration-time profile from time zero to time tau, the dosing interval, where tau=168 hours.
Time Frame: Day 22: pre-dose and 1, 6, 9, 24 and 72 hours post dose
Population: PK parameter analysis population included all enrolled participants who were treated and had at least 1 of the PK parameters of interest. Here 'Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per hour (mL/hr)
Arm/Group | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 13 | 13 | 12 | 14
milliliter per hour (mL/hr) | 28.98 (19) | 18.26 (21) | 17.59 (26) | 14.05 (15)

13. Secondary Outcome: Volume of Distribution at Steady State (Vss) of PF-04950615
Description: Vss was calculated as CL*MRT. CL was calculated as Dose/AUCtau, where AUCtau was area under the concentration-time profile from time zero to time tau (τ), the dosing interval, where tau=168 hours. MRT was mean residence time (predicted) extrapolated to infinity.
Time Frame: Day 22: pre-dose and 1, 6, 9, 24 and 72 hours post dose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter (mL)
Arm/Group | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 13 | 13 | 12 | 14
milliliter (mL) | 3815 (111) | 3221 (20) | 4035 (19) | 5285 (25)

14. Secondary Outcome: Accumulation Ratio (Rac) of PF-04950615
Description: Rac was calculated as Day 22 AUCtau divided by Day 1 AUCtau, where AUCtau is area under the concentration-time profile from time zero to time tau (τ), the dosing interval, where tau =168 hours.
Time Frame: Day 22: pre-dose and 1, 6, 9, 24 and 72 hours post dose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 13 | 13 | 12 | 14
ratio | 1.261 (12) | 1.685 (11) | 1.771 (16) | 1.964 (9)

15. Secondary Outcome: Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Day 8, 15, 22, 29 and 78
Time Frame: Baseline, Day 8, 15, 22, 29 and 78
Population: Pharmacodynamic analysis population included all enrolled participants who received at least 1 dose of study medication and had atleast 1 pharmacodynamic parameter. Here 'n' signifies those participants who were evaluable at the specified time points for each reporting group, respectively.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
milligram per deciliter (mg/dL)
  Baseline | 160.96 (19.447) | 155.04 (18.501) | 160.39 (27.326) | 155.62 (23.393) | 164.00 (21.729)
  Change at Day 8: number analyzed (Participants) | 11 | 14 | 13 | 13 | 13
  Change at Day 8 | -6.59 (11.258) | -58.89 (16.313) | -49.08 (12.708) | -68.54 (27.477) | -67.96 (27.754)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -8.21 (20.192) | -77.96 (22.181) | -70.38 (25.583) | -93.25 (31.287) | -93.79 (23.841)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -8.96 (21.416) | -84.81 (17.345) | -91.69 (20.718) | -101.92 (26.974) | -102.21 (27.277)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -13.71 (17.240) | -82.50 (20.848) | -88.00 (25.267) | -104.33 (35.026) | -104.21 (26.207)
  Change at Day 78: number analyzed (Participants) | 11 | 13 | 13 | 11 | 14
  Change at Day 78 | -4.36 (21.969) | -9.73 (19.796) | -10.15 (14.174) | -14.09 (38.162) | -65.14 (39.500)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 8: Analysis was performed using the analysis of covariance (ANCOVA) treatment, screening LDL-C stratum, study day, treatment-by-LDL-C stratum, and study day by treatment interaction as fixed effects, baseline as a covariate and participant as a random effect; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Square (LS) Mean Difference = -54.68, 95% CI 2-sided [-71.37 to -37.99], Standard Error of Mean 8.323
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; Day 8: Analysis was performed using the ANCOVA treatment, screening LDL-C stratum, study day, treatment-by-LDL-C stratum, and study day by treatment interaction as fixed effects, baseline as a covariate and participant as a random effect; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -44.18, 95% CI 2-sided [-61.28 to -27.08], Standard Error of Mean 8.530
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -64.44, 95% CI 2-sided [-81.35 to -47.53], Standard Error of Mean 8.433
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -61.75, 95% CI 2-sided [-78.36 to -45.15], Standard Error of Mean 8.282
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 15: Analysis was performed using the ANCOVA treatment, screening LDL-C stratum, study day, treatment-by-LDL-C stratum, and study day by treatment interaction as fixed effects, baseline as a covariate and participant as a random effect; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -72.16, 95% CI 2-sided [-92.40 to -51.92], Standard Error of Mean 10.097
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -63.89, 95% CI 2-sided [-84.59 to -43.19], Standard Error of Mean 10.328
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -88.69, 95% CI 2-sided [-109.39 to -68.00], Standard Error of Mean 10.327
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -84.65, 95% CI 2-sided [-104.76 to -64.54], Standard Error of Mean 10.028
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 22: Analysis was performed using the ANCOVA treatment, screening LDL-C stratum, study day, treatment-by-LDL-C stratum, and study day by treatment interaction as fixed effects, baseline as a covariate and participant as a random effect; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -78.47, 95% CI 2-sided [-96.22 to -60.71], Standard Error of Mean 8.854
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -84.45, 95% CI 2-sided [-102.51 to -66.40], Standard Error of Mean 8.998
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -96.08, 95% CI 2-sided [-114.12 to -78.03], Standard Error of Mean 8.994
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -92.33, 95% CI 2-sided [-109.80 to -74.86], Standard Error of Mean 8.703
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 29: Analysis was performed using the ANCOVA treatment, screening LDL-C stratum, study day, treatment-by-LDL-C stratum, and study day by treatment interaction as fixed effects, baseline as a covariate and participant as a random effect; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -71.41, 95% CI 2-sided [-90.51 to -52.30], Standard Error of Mean 9.534
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -76.01, 95% CI 2-sided [-95.37 to -56.65], Standard Error of Mean 9.659
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -93.78, 95% CI 2-sided [-113.18 to -74.38], Standard Error of Mean 9.678
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -89.58, 95% CI 2-sided [-108.35 to -70.81], Standard Error of Mean 9.362

16. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Day 8, 15, 22, 29 and 78
Time Frame: Day 8, 15, 22, 29 and 78
Population: Pharmacodynamic analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 pharmacodynamic parameter. Here 'n' signifies those participants who were evaluable at the specified time points for each reporting group, respectively.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
percent change
  Change at Day 8: number analyzed (Participants) | 11 | 14 | 13 | 13 | 13
  Change at Day 8 | -4.15 (6.983) | -38.53 (11.399) | -31.59 (10.032) | -44.24 (17.213) | -40.72 (14.210)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -4.39 (12.713) | -50.68 (14.566) | -45.47 (17.016) | -59.42 (19.934) | -58.02 (16.265)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -4.94 (12.826) | -54.66 (9.140) | -58.12 (13.891) | -64.59 (13.826) | -62.78 (16.665)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -8.72 (11.074) | -52.96 (11.416) | -55.25 (15.133) | -65.50 (17.327) | -63.85 (14.416)
  Change at Day 78: number analyzed (Participants) | 11 | 13 | 13 | 11 | 14
  Change at Day 78 | -2.97 (13.710) | -5.87 (12.391) | -6.50 (9.229) | -6.94 (22.385) | -40.47 (25.797)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -33.82, 95% CI 2-sided [-43.99 to -23.65], Standard Error of Mean 5.077
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -27.93, 95% CI 2-sided [-38.35 to -17.51], Standard Error of Mean 5.202
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -39.59, 95% CI 2-sided [-49.89 to -29.28], Standard Error of Mean 5.143
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -37.63, 95% CI 2-sided [-47.75 to -27.51], Standard Error of Mean 5.051
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -45.99, 95% CI 2-sided [-58.78 to -33.20], Standard Error of Mean 6.384
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -41.82, 95% CI 2-sided [-54.90 to -28.74], Standard Error of Mean 6.527
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 15: Analysis was performed using ANCOVA treatment, screening LDL-C stratum, study day, treatment-by-LDL-C stratum, and study day by treatment interaction as fixed effects, baseline as a covariate and participant as a random effect; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -56.35, 95% CI 2-sided [-69.43 to -43.27], Standard Error of Mean 6.531
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -53.45, 95% CI 2-sided [-66.17 to -40.74], Standard Error of Mean 6.344
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -49.67, 95% CI 2-sided [-60.70 to -38.64], Standard Error of Mean 5.498
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -53.92, 95% CI 2-sided [-65.14 to -42.70], Standard Error of Mean 5.592
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -60.60, 95% CI 2-sided [-71.81 to -49.38], Standard Error of Mean 5.590
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -57.67, 95% CI 2-sided [-68.53 to -46.80], Standard Error of Mean 5.413
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -44.18, 95% CI 2-sided [-55.80 to -32.57], Standard Error of Mean 5.800
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -47.28, 95% CI 2-sided [-59.06 to -35.50], Standard Error of Mean 5.881
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -57.73, 95% CI 2-sided [-69.53 to -45.94], Standard Error of Mean 5.891
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -54.96, 95% CI 2-sided [-66.38 to -43.54], Standard Error of Mean 5.701

17. Secondary Outcome: Number of Participants Achieving LDL-C Less Than (<) 70 Milligram Per Deciliter (mg/dL)
Time Frame: Day 15, 22, 29 and 36
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
Participants
  Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Day 15 | 0 | 6 | 3 | 7 | 8
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 0 | 8 | 8 | 8 | 10
  Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 29 | 0 | 6 | 6 | 9 | 10
  Day 36: number analyzed (Participants) | 11 | 13 | 13 | 12 | 13
  Day 36 | 0 | 0 | 7 | 8 | 8
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 15: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0472, Regression, Logistic; Odds Ratio (OR) = 24.972, 95% CI 2-sided [1.04 to 599.65]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; Day 15: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.1368, Regression, Logistic; Odds Ratio (OR) = 11.815, 95% CI 2-sided [0.46 to 305.54]
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 15: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0190, Regression, Logistic; Odds Ratio (OR) = 47.527, 95% CI 2-sided [1.89 to 1198.29]
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; Day 15: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0192, Regression, Logistic; Odds Ratio (OR) = 45.328, 95% CI 2-sided [1.86 to 1103.73]
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 22: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0105, Regression, Logistic; Odds Ratio (OR) = 74.273, 95% CI 2-sided [2.74 to 2014.67]
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; Day 22: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0086, Regression, Logistic; Odds Ratio (OR) = 86.088, 95% CI 2-sided [3.10 to 2389.27]
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 22: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0084, Regression, Logistic; Odds Ratio (OR) = 87.733, 95% CI 2-sided [3.14 to 2449.11]
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; Day 22: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0053, Regression, Logistic; Odds Ratio (OR) = 112.272, 95% CI 2-sided [4.07 to 3097.22]
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 29: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0403, Regression, Logistic; Odds Ratio (OR) = 27.697, 95% CI 2-sided [1.16 to 662.20]
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; Day 29: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0361, Regression, Logistic; Odds Ratio (OR) = 30.247, 95% CI 2-sided [1.25 to 733.32]
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 29: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0069, Regression, Logistic; Odds Ratio (OR) = 89.341, 95% CI 2-sided [3.43 to 2326.44]
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; Day 29: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0081, Regression, Logistic; Odds Ratio (OR) = 76.034, 95% CI 2-sided [3.08 to 1875.15]
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 36: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.9931, Regression, Logistic; Odds Ratio (OR) = 1.018, 95% CI 2-sided [0.02 to 64.41]
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; Day 36: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0259, Regression, Logistic; Odds Ratio (OR) = 38.943, 95% CI 2-sided [1.55 to 975.84]
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 36: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0142, Regression, Logistic; Odds Ratio (OR) = 57.766, 95% CI 2-sided [2.26 to 1477.88]
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; Day 36: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0179, Regression, Logistic; Odds Ratio (OR) = 48.734, 95% CI 2-sided [1.95 to 1216.90]

18. Secondary Outcome: Number of Participants Achieving LDL-C Less Than (<) 100 Milligram Per Deciliter (mg/dL)
Time Frame: Day 15, 22, 29 and 36
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
Participants
  Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Day 15 | 0 | 13 | 10 | 11 | 12
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 0 | 12 | 11 | 12 | 12
  Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 29 | 0 | 12 | 11 | 12 | 13
  Day 36: number analyzed (Participants) | 11 | 13 | 13 | 12 | 13
  Day 36 | 0 | 2 | 11 | 12 | 12
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 15: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0013, Regression, Logistic; Odds Ratio (OR) = 353.058, 95% CI 2-sided [9.95 to 12528.19]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; Day 15: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0047, Regression, Logistic; Odds Ratio (OR) = 129.984, 95% CI 2-sided [4.44 to 3808.21]
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 15: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0018, Regression, Logistic; Odds Ratio (OR) = 300.099, 95% CI 2-sided [8.35 to 10787.45]
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; Day 15: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0025, Regression, Logistic; Odds Ratio (OR) = 190.835, 95% CI 2-sided [6.34 to 5743.12]
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 22: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0018, Regression, Logistic; Odds Ratio (OR) = 255.421, 95% CI 2-sided [7.87 to 8290.22]
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; Day 22: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0034, Regression, Logistic; Odds Ratio (OR) = 150.547, 95% CI 2-sided [5.28 to 4291.89]
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 22: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0018, Regression, Logistic; Odds Ratio (OR) = 745.542, 95% CI 2-sided [11.60 to 47929.45]
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; Day 22: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0031, Regression, Logistic; Odds Ratio (OR) = 146.296, 95% CI 2-sided [5.40 to 3963.01]
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 29: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 213.512, 95% CI 2-sided [7.13 to 6396.64]
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; Day 29: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0038, Regression, Logistic; Odds Ratio (OR) = 124.439, 95% CI 2-sided [4.73 to 3277.13]
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 29: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 622.309, 95% CI 2-sided [10.51 to 36846.03]
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; Day 29: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0017, Regression, Logistic; Odds Ratio (OR) = 224.427, 95% CI 2-sided [7.63 to 6598.00]
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 36: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.2751, Regression, Logistic; Odds Ratio (OR) = 6.158, 95% CI 2-sided [0.24 to 161.08]
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; Day 36: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0038, Regression, Logistic; Odds Ratio (OR) = 152.977, 95% CI 2-sided [5.05 to 4633.92]
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 36: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 756.203, 95% CI 2-sided [11.18 to 51133.53]
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; Day 36: Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0021, Regression, Logistic; Odds Ratio (OR) = 258.938, 95% CI 2-sided [7.53 to 8902.61]

19. Secondary Outcome: Number of Participants With Greater Than or Equal to (>=) 50 Percent (%) Reduction in LDL-C From Baseline
Time Frame: Baseline, Day 15, 22, 29 and 36
Population: Pharmacodynamic analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 pharmacodynamic parameter. Here 'Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
Participants | 0 | 0 | 5 | 8 | 8
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.9580, Regression, Logistic; Odds Ratio (OR) = 0.896, 95% CI 2-sided [0.02 to 52.79]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0732, Regression, Logistic; Odds Ratio (OR) = 17.375, 95% CI 2-sided [0.76 to 394.65]
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0159, Regression, Logistic; Odds Ratio (OR) = 47.860, 95% CI 2-sided [2.07 to 1109.11]
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; Logistic regression model with treatment and baseline LDL-C stratum as factors was used for the analysis; Test type: Superiority or Other; p = 0.0264, Regression, Logistic; Odds Ratio (OR) = 33.246, 95% CI 2-sided [1.51 to 733.62]

20. Secondary Outcome: Change From Baseline in Lipid Parameters: Apolipoprotein A1 (ApoA1) at Day 8, 15, 22, 29 and 78
Time Frame: Baseline, Day 8, 15, 22, 29 and 78
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
mg/dL
  Baseline | 142.67 (20.328) | 144.43 (20.562) | 150.39 (20.863) | 143.46 (25.005) | 156.39 (28.988)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -4.00 (16.065) | 1.86 (9.698) | 0.88 (13.167) | -1.38 (10.776) | -1.75 (15.074)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -1.00 (14.918) | 13.86 (14.032) | 8.96 (13.120) | 6.83 (13.997) | 8.82 (21.116)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -5.50 (12.395) | 5.12 (13.477) | 2.27 (15.869) | -3.42 (10.025) | 6.32 (13.546)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -4.58 (12.817) | 7.96 (12.365) | 2.81 (12.377) | 1.67 (10.614) | 3.68 (16.505)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -8.92 (11.057) | -8.81 (24.972) | -6.35 (13.842) | -5.42 (15.639) | 2.46 (15.163)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.2883, ANCOVA; LS Mean Difference = 5.50, 95% CI 2-sided [-4.77 to 15.77], Standard Error of Mean 5.131
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.2563, ANCOVA; LS Mean Difference = 6.05, 95% CI 2-sided [-4.51 to 16.61], Standard Error of Mean 5.277
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.7149, ANCOVA; LS Mean Difference = 1.92, 95% CI 2-sided [-8.54 to 12.37], Standard Error of Mean 5.225
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.4480, ANCOVA; LS Mean Difference = 3.95, 95% CI 2-sided [-6.40 to 14.30], Standard Error of Mean 5.174
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0231, ANCOVA; LS Mean Difference = 14.50, 95% CI 2-sided [2.06 to 26.94], Standard Error of Mean 6.214
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0858, ANCOVA; LS Mean Difference = 11.13, 95% CI 2-sided [-1.62 to 23.87], Standard Error of Mean 6.369
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.2440, ANCOVA; LS Mean Difference = 7.57, 95% CI 2-sided [-5.30 to 20.44], Standard Error of Mean 6.431
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0702, ANCOVA; LS Mean Difference = 11.52, 95% CI 2-sided [-0.98 to 24.03], Standard Error of Mean 6.249
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0531, ANCOVA; LS Mean Difference = 9.64, 95% CI 2-sided [-0.13 to 19.41], Standard Error of Mean 4.878
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0758, ANCOVA; LS Mean Difference = 8.93, 95% CI 2-sided [-0.96 to 18.83], Standard Error of Mean 4.940
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.6965, ANCOVA; LS Mean Difference = 1.95, 95% CI 2-sided [-8.01 to 11.92], Standard Error of Mean 4.975
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0071, ANCOVA; LS Mean Difference = 13.52, 95% CI 2-sided [3.83 to 23.22], Standard Error of Mean 4.842
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.0339, ANCOVA; LS Mean Difference = 11.20, 95% CI 2-sided [0.88 to 21.52], Standard Error of Mean 5.155
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.1075, ANCOVA; LS Mean Difference = 8.56, 95% CI 2-sided [-1.92 to 19.03], Standard Error of Mean 5.235
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.2601, ANCOVA; LS Mean Difference = 5.98, 95% CI 2-sided [-4.54 to 16.50], Standard Error of Mean 5.258
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.0570, ANCOVA; LS Mean Difference = 9.96, 95% CI 2-sided [-0.31 to 20.24], Standard Error of Mean 5.132

21. Secondary Outcome: Change From Baseline in Lipid Parameters: Apolipoprotein B (ApoB) at Day 8, 15, 22, 29 and 78
Time Frame: Baseline, Day 8, 15, 22, 29 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
mg/dL
  Baseline | 126.54 (13.662) | 124.04 (16.454) | 120.32 (16.199) | 125.62 (18.377) | 119.57 (16.804)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -7.79 (15.901) | -38.39 (8.150) | -32.69 (11.479) | -46.46 (17.016) | -41.36 (12.796)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -9.21 (10.279) | -49.11 (15.713) | -46.00 (19.321) | -61.83 (22.850) | -56.29 (14.567)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -7.21 (12.520) | -52.54 (13.124) | -52.38 (14.826) | -65.17 (21.560) | -59.44 (19.275)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -8.46 (12.945) | -55.54 (14.941) | -54.08 (14.850) | -70.75 (25.561) | -63.66 (16.555)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -8.29 (12.894) | -8.46 (18.284) | -9.38 (13.489) | -11.92 (17.403) | -39.36 (19.171)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -32.88, 95% CI 2-sided [-42.93 to -22.84], Standard Error of Mean 5.008
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -30.80, 95% CI 2-sided [-41.34 to -20.26], Standard Error of Mean 5.260
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -39.98, 95% CI 2-sided [-50.18 to -29.77], Standard Error of Mean 5.088
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -38.37, 95% CI 2-sided [-48.54 to -28.20], Standard Error of Mean 5.070
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -42.18, 95% CI 2-sided [-54.73 to -29.63], Standard Error of Mean 6.271
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -42.69, 95% CI 2-sided [-55.72 to -29.67], Standard Error of Mean 6.512
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -54.56, 95% CI 2-sided [-67.45 to -41.67], Standard Error of Mean 6.445
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -51.89, 95% CI 2-sided [-64.54 to -39.25], Standard Error of Mean 6.321
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 95, ANCOVA; LS Mean Difference = -47.35, 95% CI 2-sided [-58.10 to -36.59], Standard Error of Mean 5.359
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -51.08, 95% CI 2-sided [-62.24 to -39.91], Standard Error of Mean 5.566
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -59.89, 95% CI 2-sided [-70.89 to -48.89], Standard Error of Mean 5.482
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -57.03, 95% CI 2-sided [-67.83 to -46.24], Standard Error of Mean 5.377
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -49.06, 95% CI 2-sided [-60.61 to -37.51], Standard Error of Mean 5.767
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -51.52, 95% CI 2-sided [-63.48 to -39.56], Standard Error of Mean 5.974
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -64.22, 95% CI 2-sided [-76.04 to -52.40], Standard Error of Mean 5.901
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -60.01, 95% CI 2-sided [-71.59 to -48.42], Standard Error of Mean 5.785

22. Secondary Outcome: Change From Baseline in Lipid Parameters: Total Cholesterol at Day 8, 15, 22, 29 and 78
Time Frame: Baseline, Day 8, 15, 22, 29 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
mg/dL
  Baseline | 237.75 (24.940) | 233.21 (26.471) | 239.36 (32.827) | 242.54 (31.408) | 247.21 (24.410)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -8.67 (12.841) | -61.29 (18.605) | -51.96 (18.394) | -77.15 (28.981) | -71.50 (28.657)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -11.33 (23.714) | -77.43 (22.270) | -70.96 (30.673) | -97.67 (35.386) | -94.79 (24.196)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -7.58 (24.265) | -85.00 (21.184) | -89.81 (23.173) | -112.08 (36.393) | -100.14 (26.658)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -14.67 (17.127) | -83.46 (23.107) | -88.35 (26.534) | -116.75 (46.591) | -104.14 (26.623)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -1.25 (19.760) | -11.38 (31.685) | -11.88 (20.431) | -16.42 (35.522) | -63.64 (40.832)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -54.91, 95% CI 2-sided [-75.54 to -34.29], Standard Error of Mean 10.392
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -44.07, 95% CI 2-sided [-65.21 to -22.94], Standard Error of Mean 10.646
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -67.98, 95% CI 2-sided [-88.92 to -47.05], Standard Error of Mean 10.547
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -60.51, 95% CI 2-sided [-81.11 to -39.90], Standard Error of Mean 10.381
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -68.39, 95% CI 2-sided [-89.02 to -47.76], Standard Error of Mean 10.392
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -60.41, 95% CI 2-sided [-81.54 to -39.27], Standard Error of Mean 10.646
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -86.60, 95% CI 2-sided [-107.74 to -65.46], Standard Error of Mean 10.656
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -81.13, 95% CI 2-sided [-101.73 to -60.52], Standard Error of Mean 10.381
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -80.16, 95% CI 2-sided [-100.96 to -59.37], Standard Error of Mean 10.479
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -83.00, 95% CI 2-sided [-104.14 to -61.87], Standard Error of Mean 10.646
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -104.77, 95% CI 2-sided [-125.91 to -83.62], Standard Error of Mean 10.656
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -90.23, 95% CI 2-sided [-110.84 to -69.63], Standard Error of Mean 10.381
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -71.54, 95% CI 2-sided [-92.34 to -50.75], Standard Error of Mean 10.479
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -74.46, 95% CI 2-sided [-95.59 to -53.32], Standard Error of Mean 10.646
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -102.35, 95% CI 2-sided [-123.49 to -81.21], Standard Error of Mean 10.656
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -87.15, 95% CI 2-sided [-107.76 to -66.55], Standard Error of Mean 10.381

23. Secondary Outcome: Change From Baseline in Lipid Parameters: High Density Lipoprotein Cholesterol (HDL-C) at Day 8, 15, 22, 29 and 78
Time Frame: Baseline, Day 8, 15, 22, 29 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
mg/dL
  Baseline | 46.29 (11.696) | 47.75 (10.864) | 52.89 (12.837) | 49.23 (14.621) | 55.64 (15.687)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -1.71 (5.211) | 0.18 (5.052) | 0.23 (3.908) | -0.92 (4.821) | 0.00 (5.349)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -2.13 (5.050) | 4.39 (5.936) | 2.23 (3.930) | 1.58 (7.141) | 2.21 (6.830)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -0.13 (4.354) | 3.31 (4.671) | 2.54 (6.280) | 0.17 (4.499) | 4.79 (7.122)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -0.46 (7.149) | 3.77 (6.559) | 2.46 (7.304) | 0.92 (7.122) | 5.36 (4.483)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -1.29 (6.315) | -1.31 (10.355) | -1.46 (4.832) | -0.25 (5.586) | 5.14 (6.443)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.3064, ANCOVA; LS Mean Difference = 2.01, 95% CI 2-sided [-1.89 to 5.90], Standard Error of Mean 1.945
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.1922, ANCOVA; LS Mean Difference = 2.67, 95% CI 2-sided [-1.38 to 6.73], Standard Error of Mean 2.025
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.6827, ANCOVA; LS Mean Difference = 0.82, 95% CI 2-sided [-3.16 to 4.79], Standard Error of Mean 1.984
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.2211, ANCOVA; LS Mean Difference = 2.45, 95% CI 2-sided [-1.52 to 6.42], Standard Error of Mean 1.981
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0033, ANCOVA; LS Mean Difference = 6.64, 95% CI 2-sided [2.31 to 10.97], Standard Error of Mean 2.158
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0269, ANCOVA; LS Mean Difference = 5.09, 95% CI 2-sided [0.60 to 9.57], Standard Error of Mean 2.237
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0890, ANCOVA; LS Mean Difference = 3.87, 95% CI 2-sided [-0.61 to 8.34], Standard Error of Mean 2.232
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0242, ANCOVA; LS Mean Difference = 5.08, 95% CI 2-sided [0.69 to 9.47], Standard Error of Mean 2.190
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.1270, ANCOVA; LS Mean Difference = 3.25, 95% CI 2-sided [-0.95 to 7.46], Standard Error of Mean 2.101
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.1199, ANCOVA; LS Mean Difference = 3.40, 95% CI 2-sided [-0.91 to 7.70], Standard Error of Mean 2.151
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.8123, ANCOVA; LS Mean Difference = 0.51, 95% CI 2-sided [-3.79 to 4.82], Standard Error of Mean 2.150
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0095, ANCOVA; LS Mean Difference = 5.65, 95% CI 2-sided [1.44 to 9.87], Standard Error of Mean 2.106
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.1141, ANCOVA; LS Mean Difference = 4.00, 95% CI 2-sided [-0.99 to 8.99], Standard Error of Mean 2.492
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.1552, ANCOVA; LS Mean Difference = 3.65, 95% CI 2-sided [-1.42 to 8.73], Standard Error of Mean 2.536
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.5407, ANCOVA; LS Mean Difference = 1.57, 95% CI 2-sided [-3.53 to 6.67], Standard Error of Mean 2.547
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.0107, ANCOVA; LS Mean Difference = 6.56, 95% CI 2-sided [1.58 to 11.53], Standard Error of Mean 2.485

24. Secondary Outcome: Change From Baseline In Lipid Parameters: Non High Density Lipoprotein Cholesterol (Non HDL-C) at Day 8, 15, 22, 29 and 78
Time Frame: Baseline, Day 8, 15, 22, 29 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
mg/dL
  Baseline | 191.46 (20.999) | 185.46 (26.890) | 186.46 (29.171) | 193.31 (34.922) | 191.57 (26.355)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -6.96 (10.212) | -61.46 (17.091) | -52.19 (16.982) | -76.23 (27.030) | -71.50 (29.506)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -9.21 (21.912) | -81.82 (22.163) | -73.19 (31.471) | -99.25 (34.162) | -97.00 (25.070)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -7.46 (24.362) | -88.31 (20.754) | -92.35 (21.685) | -112.25 (35.962) | -104.93 (28.080)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -14.21 (13.327) | -87.23 (19.842) | -90.81 (25.136) | -117.67 (45.816) | -109.50 (28.156)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | 0.04 (22.738) | -10.08 (28.522) | -10.42 (19.339) | -16.17 (33.701) | -68.79 (43.324)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -60.35, 95% CI 2-sided [-76.74 to -43.97], Standard Error of Mean 8.152
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -52.53, 95% CI 2-sided [-69.45 to -35.61], Standard Error of Mean 8.422
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -69.46, 95% CI 2-sided [-86.06 to -52.86], Standard Error of Mean 8.260
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -66.25, 95% CI 2-sided [-82.55 to -49.94], Standard Error of Mean 8.112
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -78.46, 95% CI 2-sided [-100.05 to -56.87], Standard Error of Mean 10.766
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -71.28, 95% CI 2-sided [-93.43 to -49.13], Standard Error of Mean 11.051
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -91.83, 95% CI 2-sided [-113.92 to -69.74], Standard Error of Mean 11.018
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -89.50, 95% CI 2-sided [-111.03 to -67.97], Standard Error of Mean 10.736
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -86.73, 95% CI 2-sided [-103.73 to -69.72], Standard Error of Mean 8.452
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -92.18, 95% CI 2-sided [-109.57 to -74.80], Standard Error of Mean 8.643
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -106.06, 95% CI 2-sided [-123.34 to -88.78], Standard Error of Mean 8.585
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -99.18, 95% CI 2-sided [-115.95 to -82.40], Standard Error of Mean 8.334
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -79.07, 95% CI 2-sided [-96.22 to -61.93], Standard Error of Mean 8.557
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -83.89, 95% CI 2-sided [-101.40 to -66.39], Standard Error of Mean 8.736
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -104.74, 95% CI 2-sided [-122.13 to -87.35], Standard Error of Mean 8.679
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -97.00, 95% CI 2-sided [-113.89 to -80.11], Standard Error of Mean 8.426

25. Secondary Outcome: Change From Baseline In Lipid Parameters: Triglycerides (TG) at Day 8, 15, 22, 29 and 78
Time Frame: Baseline, Day 8, 15, 22, 29 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
mg/dL
  Baseline | 152.92 (52.761) | 152.00 (55.166) | 130.36 (41.199) | 182.27 (117.963) | 137.96 (70.799)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | 4.33 (53.163) | -12.21 (52.707) | -15.69 (41.689) | -32.35 (52.814) | -2.18 (66.044)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -4.92 (47.001) | -19.00 (32.268) | -13.92 (44.051) | -23.54 (40.176) | -16.32 (32.999)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | 7.75 (39.352) | -17.62 (45.629) | -3.54 (39.199) | -45.29 (82.959) | -13.75 (47.976)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -3.00 (43.389) | -24.23 (36.103) | -14.38 (53.705) | -60.21 (102.224) | -26.25 (29.632)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | 52.33 (177.350) | -1.77 (52.488) | -1.00 (35.576) | 12.21 (108.874) | -18.25 (40.930)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.4480, ANCOVA; LS Mean Difference = -22.30, 95% CI 2-sided [-80.08 to 35.49], Standard Error of Mean 29.336
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.2809, ANCOVA; LS Mean Difference = -32.52, 95% CI 2-sided [-91.80 to 26.76], Standard Error of Mean 30.091
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.2875, ANCOVA; LS Mean Difference = -31.92, 95% CI 2-sided [-90.90 to 27.07], Standard Error of Mean 29.942
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.5743, ANCOVA; LS Mean Difference = -16.52, 95% CI 2-sided [-74.38 to 41.33], Standard Error of Mean 29.370
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.4997, ANCOVA; LS Mean Difference = -19.83, 95% CI 2-sided [-77.62 to 37.96], Standard Error of Mean 29.336
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.4756, ANCOVA; LS Mean Difference = -21.50, 95% CI 2-sided [-80.78 to 37.78], Standard Error of Mean 30.091
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.5610, ANCOVA; LS Mean Difference = -17.73, 95% CI 2-sided [-77.73 to 42.26], Standard Error of Mean 30.458
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.4667, ANCOVA; LS Mean Difference = -21.41, 95% CI 2-sided [-79.27 to 36.44], Standard Error of Mean 29.370
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.3045, ANCOVA; LS Mean Difference = -30.70, 95% CI 2-sided [-89.45 to 28.06], Standard Error of Mean 29.828
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.4301, ANCOVA; LS Mean Difference = -23.78, 95% CI 2-sided [-83.06 to 35.50], Standard Error of Mean 30.091
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0881, ANCOVA; LS Mean Difference = -52.15, 95% CI 2-sided [-112.15 to 7.85], Standard Error of Mean 30.458
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.2844, ANCOVA; LS Mean Difference = -31.51, 95% CI 2-sided [-89.36 to 26.35], Standard Error of Mean 29.370
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.3741, ANCOVA; LS Mean Difference = -26.56, 95% CI 2-sided [-85.32 to 32.19], Standard Error of Mean 29.828
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.4283, ANCOVA; LS Mean Difference = -23.88, 95% CI 2-sided [-83.16 to 35.40], Standard Error of Mean 30.091
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.0657, ANCOVA; LS Mean Difference = -56.32, 95% CI 2-sided [-116.31 to 3.68], Standard Error of Mean 30.458
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.2586, ANCOVA; LS Mean Difference = -33.26, 95% CI 2-sided [-91.11 to 24.60], Standard Error of Mean 29.370

26. Secondary Outcome: Percent Change From Baseline in Lipid Parameters: Apolipoprotein A1 (ApoA1) at Day 8, 15, 22, 29 and 78
Time Frame: Day 8, 15, 22, 29 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
percent change
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -2.15 (10.895) | 1.38 (6.508) | 0.55 (8.065) | -1.17 (7.549) | -0.19 (9.462)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -0.18 (10.362) | 10.03 (10.615) | 5.67 (8.409) | 4.99 (9.450) | 6.11 (14.252)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -3.38 (8.315) | 4.01 (9.735) | 1.90 (10.085) | -1.61 (6.994) | 4.92 (9.366)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -2.62 (8.538) | 5.82 (8.244) | 1.80 (8.623) | 1.20 (7.435) | 3.51 (11.179)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -5.85 (7.270) | -4.61 (15.035) | -3.48 (9.082) | -3.77 (10.868) | 3.20 (11.505)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.3326, ANCOVA; LS Mean Difference = 3.33, 95% CI 2-sided [-3.49 to 10.14], Standard Error of Mean 3.404
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.2967, ANCOVA; LS Mean Difference = 3.69, 95% CI 2-sided [-3.32 to 10.70], Standard Error of Mean 3.502
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.8812, ANCOVA; LS Mean Difference = 0.52, 95% CI 2-sided [-6.42 to 7.46], Standard Error of Mean 3.466
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.3227, ANCOVA; LS Mean Difference = 3.42, 95% CI 2-sided [-3.45 to 10.30], Standard Error of Mean 3.433
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0210, ANCOVA; LS Mean Difference = 10.01, 95% CI 2-sided [1.56 to 18.46], Standard Error of Mean 4.221
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.1192, ANCOVA; LS Mean Difference = 6.84, 95% CI 2-sided [-1.82 to 15.49], Standard Error of Mean 4.326
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.2529, ANCOVA; LS Mean Difference = 5.04, 95% CI 2-sided [-3.69 to 13.78], Standard Error of Mean 4.367
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0725, ANCOVA; LS Mean Difference = 7.76, 95% CI 2-sided [-0.73 to 16.25], Standard Error of Mean 4.244
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0405, ANCOVA; LS Mean Difference = 6.74, 95% CI 2-sided [0.30 to 13.18], Standard Error of Mean 3.214
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0593, ANCOVA; LS Mean Difference = 6.27, 95% CI 2-sided [-0.25 to 12.80], Standard Error of Mean 3.258
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.5936, ANCOVA; LS Mean Difference = 1.76, 95% CI 2-sided [-4.81 to 8.33], Standard Error of Mean 3.279
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0034, ANCOVA; LS Mean Difference = 9.78, 95% CI 2-sided [3.38 to 16.17], Standard Error of Mean 3.192
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.0305, ANCOVA; LS Mean Difference = 7.60, 95% CI 2-sided [0.74 to 14.46], Standard Error of Mean 3.428
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.1252, ANCOVA; LS Mean Difference = 5.41, 95% CI 2-sided [-1.55 to 12.37], Standard Error of Mean 3.479
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.2923, ANCOVA; LS Mean Difference = 3.71, 95% CI 2-sided [-3.28 to 10.71], Standard Error of Mean 3.495
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.0297, ANCOVA; LS Mean Difference = 7.60, 95% CI 2-sided [0.78 to 14.43], Standard Error of Mean 3.411

27. Secondary Outcome: Percent Change From Baseline In Lipid Parameters: Apolipoprotein B (ApoB) at Day 8, 15, 22, 29 and 78
Time Frame: Day 8, 15, 22, 29 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
percent change
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -5.78 (12.548) | -31.37 (7.019) | -27.78 (9.784) | -36.61 (12.248) | -34.71 (9.872)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -7.08 (7.974) | -39.63 (11.339) | -38.94 (15.373) | -49.03 (15.663) | -47.45 (12.424)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -5.17 (9.548) | -42.06 (8.865) | -43.87 (10.909) | -51.52 (12.657) | -49.45 (13.498)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -6.61 (10.206) | -44.37 (10.311) | -45.51 (12.176) | -55.74 (15.477) | -53.15 (10.682)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -6.24 (10.119) | -6.11 (13.750) | -7.95 (11.527) | -8.40 (13.819) | -33.66 (17.828)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -26.35, 95% CI 2-sided [-34.59 to -18.10], Standard Error of Mean 4.117
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -24.29, 95% CI 2-sided [-32.95 to -15.63], Standard Error of Mean 4.325
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -31.20, 95% CI 2-sided [-39.58 to -22.83], Standard Error of Mean 4.182
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -30.43, 95% CI 2-sided [-38.78 to -22.08], Standard Error of Mean 4.169
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -33.30, 95% CI 2-sided [-43.42 to -23.19], Standard Error of Mean 5.055
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -34.14, 95% CI 2-sided [-44.65 to -23.63], Standard Error of Mean 5.255
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -42.57, 95% CI 2-sided [-52.96 to -32.18], Standard Error of Mean 5.194
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -41.87, 95% CI 2-sided [-52.07 to -31.67], Standard Error of Mean 5.097
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -37.75, 95% CI 2-sided [-46.46 to -29.05], Standard Error of Mean 4.343
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -40.98, 95% CI 2-sided [-50.04 to -31.93], Standard Error of Mean 4.519
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -46.98, 95% CI 2-sided [-55.88 to -38.08], Standard Error of Mean 4.441
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -45.77, 95% CI 2-sided [-54.52 to -37.03], Standard Error of Mean 4.363
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -38.61, 95% CI 2-sided [-47.85 to -29.37], Standard Error of Mean 4.616
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -41.19, 95% CI 2-sided [-50.78 to -31.60], Standard Error of Mean 4.795
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -49.75, 95% CI 2-sided [-59.20 to -40.30], Standard Error of Mean 4.722
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -48.04, 95% CI 2-sided [-57.33 to -38.76], Standard Error of Mean 4.639

28. Secondary Outcome: Percent Change From Baseline In Lipid Parameters: Total Cholesterol at Day 8, 15, 22, 29 and 78
Time Frame: Day 8, 15, 22, 29 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
percent change
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -3.73 (5.594) | -26.43 (7.582) | -22.11 (8.292) | -31.68 (11.543) | -28.70 (10.002)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -4.46 (10.151) | -33.35 (9.238) | -30.59 (13.208) | -39.69 (13.307) | -38.77 (10.906)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -2.61 (9.708) | -36.44 (7.736) | -37.81 (9.438) | -45.23 (11.101) | -40.69 (10.542)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -6.12 (7.275) | -35.76 (8.855) | -37.12 (11.045) | -46.81 (15.606) | -42.24 (9.692)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -0.90 (8.320) | -4.28 (13.040) | -5.11 (8.907) | -5.49 (14.026) | -26.16 (17.561)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -22.70, 95% CI 2-sided [-31.06 to -14.34], Standard Error of Mean 4.211
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -18.60, 95% CI 2-sided [-27.17 to -10.03], Standard Error of Mean 4.315
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -27.97, 95% CI 2-sided [-36.46 to -19.49], Standard Error of Mean 4.274
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -24.89, 95% CI 2-sided [-33.24 to -16.54], Standard Error of Mean 4.207
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -28.89, 95% CI 2-sided [-37.25 to -20.53], Standard Error of Mean 4.211
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -26.35, 95% CI 2-sided [-34.92 to -17.79], Standard Error of Mean 4.315
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -35.89, 95% CI 2-sided [-44.46 to -27.33], Standard Error of Mean 4.318
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -34.23, 95% CI 2-sided [-42.58 to -25.88], Standard Error of Mean 4.207
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -33.96, 95% CI 2-sided [-42.39 to -25.53], Standard Error of Mean 4.246
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -35.41, 95% CI 2-sided [-43.98 to -26.85], Standard Error of Mean 4.315
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -43.28, 95% CI 2-sided [-51.85 to -34.71], Standard Error of Mean 4.318
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -38.00, 95% CI 2-sided [-46.35 to -29.65], Standard Error of Mean 4.207
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -29.77, 95% CI 2-sided [-38.19 to -21.34], Standard Error of Mean 4.246
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -31.22, 95% CI 2-sided [-39.79 to -22.65], Standard Error of Mean 4.315
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -41.34, 95% CI 2-sided [-49.91 to -32.78], Standard Error of Mean 4.318
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -36.04, 95% CI 2-sided [-44.39 to -27.69], Standard Error of Mean 4.207

29. Secondary Outcome: Percent Change From Baseline In Lipid Parameters: High Density Lipoprotein Cholesterol (HDL-C) at Day 8, 15, 22, 29 and 78
Time Frame: Day 8, 15, 22, 29 and 78
Population: Pharmacodynamic analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 pharmacodynamic parameter.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
percent change
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -2.75 (11.363) | 1.26 (10.469) | 0.31 (7.401) | -2.64 (9.055) | 0.61 (10.217)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -3.98 (10.134) | 10.54 (14.406) | 4.72 (8.025) | 4.39 (11.643) | 5.56 (13.089)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | 0.48 (9.693) | 8.01 (10.268) | 5.49 (11.126) | 1.78 (9.431) | 9.83 (14.119)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | 0.02 (14.389) | 9.02 (14.218) | 4.55 (12.030) | 3.56 (12.870) | 11.44 (10.270)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -1.40 (13.662) | 0.24 (19.628) | -2.24 (8.900) | -2.32 (11.310) | 11.35 (13.124)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.2690, ANCOVA; LS Mean Difference = 4.44, 95% CI 2-sided [-3.53 to 12.41], Standard Error of Mean 3.975
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.2122, ANCOVA; LS Mean Difference = 5.22, 95% CI 2-sided [-3.07 to 13.50], Standard Error of Mean 4.133
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.8953, ANCOVA; LS Mean Difference = 0.54, 95% CI 2-sided [-7.59 to 8.67], Standard Error of Mean 4.054
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.1723, ANCOVA; LS Mean Difference = 5.59, 95% CI 2-sided [-2.51 to 13.70], Standard Error of Mean 4.045
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0010, ANCOVA; LS Mean Difference = 14.95, 95% CI 2-sided [6.34 to 23.56], Standard Error of Mean 4.293
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0179, ANCOVA; LS Mean Difference = 10.86, 95% CI 2-sided [1.95 to 19.78], Standard Error of Mean 4.451
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0462, ANCOVA; LS Mean Difference = 9.06, 95% CI 2-sided [0.16 to 17.96], Standard Error of Mean 4.440
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.0091, ANCOVA; LS Mean Difference = 11.78, 95% CI 2-sided [3.05 to 20.52], Standard Error of Mean 4.358
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0774, ANCOVA; LS Mean Difference = 7.31, 95% CI 2-sided [-0.83 to 15.45], Standard Error of Mean 4.064
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0909, ANCOVA; LS Mean Difference = 7.16, 95% CI 2-sided [-1.18 to 15.50], Standard Error of Mean 4.165
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.6107, ANCOVA; LS Mean Difference = 2.13, 95% CI 2-sided [-6.20 to 10.45], Standard Error of Mean 4.157
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.0062, ANCOVA; LS Mean Difference = 11.59, 95% CI 2-sided [3.42 to 19.75], Standard Error of Mean 4.076
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.0702, ANCOVA; LS Mean Difference = 8.69, 95% CI 2-sided [-0.74 to 18.13], Standard Error of Mean 4.712
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.1692, ANCOVA; LS Mean Difference = 6.69, 95% CI 2-sided [-2.93 to 16.32], Standard Error of Mean 4.807
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.3751, ANCOVA; LS Mean Difference = 4.31, 95% CI 2-sided [-5.34 to 13.96], Standard Error of Mean 4.819
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.0053, ANCOVA; LS Mean Difference = 13.65, 95% CI 2-sided [4.23 to 23.08], Standard Error of Mean 4.709

30. Secondary Outcome: Percent Change From Baseline In Lipid Parameters: Non High Density Lipoprotein Cholesterol (Non HDL-C) at Day 8, 15, 22, 29 and 78
Time Frame: Day 8, 15, 22, 29 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
percent change
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -3.85 (5.557) | -33.32 (8.161) | -28.56 (8.868) | -39.11 (12.195) | -36.85 (11.918)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -4.33 (11.789) | -44.54 (12.261) | -40.54 (15.915) | -50.81 (14.320) | -50.85 (12.789)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -3.27 (12.091) | -47.43 (7.666) | -50.15 (10.327) | -57.08 (10.801) | -54.61 (11.948)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -7.45 (7.261) | -46.96 (8.425) | -49.29 (12.890) | -59.12 (15.643) | -56.98 (10.994)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -0.13 (11.797) | -4.84 (14.681) | -5.97 (10.711) | -6.62 (16.960) | -36.83 (24.401)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -30.64, 95% CI 2-sided [-38.56 to -22.72], Standard Error of Mean 3.951
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -26.62, 95% CI 2-sided [-34.80 to -18.44], Standard Error of Mean 4.084
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -35.27, 95% CI 2-sided [-43.29 to -27.24], Standard Error of Mean 4.003
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -33.42, 95% CI 2-sided [-41.30 to -25.54], Standard Error of Mean 3.931
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -41.38, 95% CI 2-sided [-52.34 to -30.42], Standard Error of Mean 5.467
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -38.12, 95% CI 2-sided [-49.36 to -26.88], Standard Error of Mean 5.610
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -47.42, 95% CI 2-sided [-58.64 to -36.20], Standard Error of Mean 5.599
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -46.93, 95% CI 2-sided [-57.87 to -36.00], Standard Error of Mean 5.453
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -45.37, 95% CI 2-sided [-53.96 to -36.77], Standard Error of Mean 4.275
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -48.78, 95% CI 2-sided [-57.58 to -39.99], Standard Error of Mean 4.374
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -54.49, 95% CI 2-sided [-63.23 to -45.75], Standard Error of Mean 4.346
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -51.75, 95% CI 2-sided [-60.25 to -43.26], Standard Error of Mean 4.222
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -40.82, 95% CI 2-sided [-49.58 to -32.07], Standard Error of Mean 4.373
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -43.75, 95% CI 2-sided [-52.68 to -34.81], Standard Error of Mean 4.464
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -52.36, 95% CI 2-sided [-61.25 to -43.48], Standard Error of Mean 4.437
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -49.94, 95% CI 2-sided [-58.58 to -41.31], Standard Error of Mean 4.312

31. Secondary Outcome: Percent Change From Baseline In Lipid Parameters: Triglycerides (TG) at Day 8, 15, 22, 29 and 78
Time Frame: Day 8, 15, 22, 29 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
percent change
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -2.25 (30.696) | 0.47 (36.664) | -9.47 (33.634) | -15.52 (25.106) | -1.90 (35.794)
  Change at Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Change at Day 15 | -1.76 (38.074) | -9.97 (19.639) | -8.88 (29.664) | -8.87 (16.916) | -8.36 (32.603)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | 5.29 (25.939) | -9.14 (24.192) | -2.82 (31.720) | -13.00 (28.724) | -8.11 (31.027)
  Change at Day 29: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 29 | -6.35 (24.168) | -15.68 (17.890) | -13.18 (39.826) | -19.81 (34.900) | -18.32 (21.062)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | 35.06 (123.074) | 4.27 (33.925) | -2.18 (32.081) | 4.74 (43.369) | -12.42 (28.128)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.9789, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-39.08 to 38.04], Standard Error of Mean 19.581
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.5525, ANCOVA; LS Mean Difference = -11.94, 95% CI 2-sided [-51.46 to 27.59], Standard Error of Mean 20.069
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.5035, ANCOVA; LS Mean Difference = -13.39, 95% CI 2-sided [-52.73 to 25.96], Standard Error of Mean 19.979
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.8302, ANCOVA; LS Mean Difference = -4.21, 95% CI 2-sided [-42.81 to 34.39], Standard Error of Mean 19.601
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.5590, ANCOVA; LS Mean Difference = -11.45, 95% CI 2-sided [-50.01 to 27.10], Standard Error of Mean 19.581
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.5558, ANCOVA; LS Mean Difference = -11.84, 95% CI 2-sided [-51.36 to 27.69], Standard Error of Mean 20.069
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.6835, ANCOVA; LS Mean Difference = -8.30, 95% CI 2-sided [-48.34 to 31.74], Standard Error of Mean 20.332
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.5699, ANCOVA; LS Mean Difference = -11.15, 95% CI 2-sided [-49.75 to 27.45], Standard Error of Mean 19.601
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.3826, ANCOVA; LS Mean Difference = -17.42, 95% CI 2-sided [-56.64 to 21.80], Standard Error of Mean 19.918
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.5233, ANCOVA; LS Mean Difference = -12.83, 95% CI 2-sided [-52.35 to 26.70], Standard Error of Mean 20.069
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.3391, ANCOVA; LS Mean Difference = -19.47, 95% CI 2-sided [-59.51 to 20.57], Standard Error of Mean 20.332
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.3606, ANCOVA; LS Mean Difference = -17.95, 95% CI 2-sided [-56.55 to 20.65], Standard Error of Mean 19.601
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.5364, ANCOVA; LS Mean Difference = -12.33, 95% CI 2-sided [-51.55 to 26.89], Standard Error of Mean 19.918
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 0.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.5651, ANCOVA; LS Mean Difference = -11.56, 95% CI 2-sided [-51.08 to 27.96], Standard Error of Mean 20.069
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 1.0 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.4719, ANCOVA; LS Mean Difference = -14.65, 95% CI 2-sided [-54.69 to 25.39], Standard Error of Mean 20.332
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 1.50 mg/kg; [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; p = 0.3999, ANCOVA; LS Mean Difference = -16.53, 95% CI 2-sided [-55.13 to 22.07], Standard Error of Mean 19.601

32. Secondary Outcome: Change From Baseline In Low Density Lipoprotein Cholesterol (LDL-C) Particle Size at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Baseline, Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nanometer (nm)
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nanometer (nm)
  Baseline | 20.37 (0.713) | 20.48 (0.833) | 21.04 (1.059) | 20.66 (1.018) | 21.18 (1.132)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | 0.00 (0.600) | 0.07 (0.334) | 0.06 (0.399) | -0.02 (0.446) | 0.09 (0.380)
  Change at Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 15 | -0.23 (0.661) | -0.13 (0.403) | 0.19 (0.463) | -0.08 (0.496) | 0.05 (0.372)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -0.05 (0.403) | 0.24 (0.333) | 0.10 (0.567) | 0.08 (0.564) | 0.08 (0.507)
  Change at Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 36 | -0.13 (0.382) | 0.01 (0.352) | 0.22 (0.518) | 0.07 (0.509) | 0.09 (0.766)
  Change at Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 50 | -0.04 (0.487) | -0.08 (0.285) | -0.18 (0.463) | -0.02 (0.327) | 0.11 (0.595)
  Change at Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 64 | -0.19 (0.601) | -0.19 (0.413) | -0.18 (0.426) | -0.08 (0.379) | 0.04 (0.497)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -0.13 (0.367) | 0.11 (0.551) | -0.15 (0.533) | -0.09 (0.323) | 0.08 (0.435)

33. Secondary Outcome: Change From Baseline In Small Low Density Lipoprotein Cholesterol (LDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Baseline, Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nanomoles per liter (nmol/L)
  Baseline | 1436.42 (476.114) | 1285.21 (510.295) | 982.14 (660.248) | 1163.69 (625.676) | 870.07 (564.004)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -104.67 (421.388) | -435.86 (323.733) | -304.85 (390.365) | -459.31 (379.905) | -321.71 (311.160)
  Change at Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 15 | -21.08 (348.697) | -521.15 (397.925) | -450.31 (458.385) | -567.67 (533.371) | -470.93 (348.889)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -62.92 (369.272) | -665.23 (392.357) | -450.85 (531.247) | -696.42 (589.692) | -513.07 (392.796)
  Change at Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 36 | -58.92 (273.321) | -245.77 (326.908) | -534.62 (480.776) | -697.50 (565.896) | -540.93 (394.389)
  Change at Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 50 | 38.58 (341.805) | 19.31 (136.299) | -88.15 (311.715) | -450.17 (475.951) | -514.64 (444.216)
  Change at Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 64 | 35.58 (410.428) | 102.15 (222.450) | 60.00 (245.038) | -165.33 (302.403) | -441.29 (420.139)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -17.25 (256.900) | -70.92 (356.896) | 39.00 (417.482) | -57.33 (364.799) | -299.43 (315.715)

34. Secondary Outcome: Change From Baseline In Medium Low Density Lipoprotein Cholesterol (LDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Baseline, Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nmol/L
  Baseline | 302.67 (103.271) | 257.57 (98.358) | 196.57 (128.296) | 237.31 (135.958) | 171.14 (114.370)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -45.33 (77.296) | -70.71 (66.675) | -52.77 (77.953) | -89.62 (96.271) | -58.00 (69.471)
  Change at Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 15 | -17.92 (90.062) | -88.15 (85.983) | -83.85 (91.519) | -105.25 (124.532) | -83.29 (70.268)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -17.33 (72.118) | -113.54 (84.567) | -77.54 (104.141) | -126.50 (134.014) | -95.93 (80.612)
  Change at Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 36 | -26.58 (70.370) | -39.85 (75.660) | -103.46 (96.958) | -128.83 (128.898) | -95.93 (75.083)
  Change at Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 50 | -7.42 (67.594) | 16.77 (46.490) | -1.23 (63.816) | -76.00 (105.963) | -89.57 (89.102)
  Change at Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 64 | -7.50 (91.363) | 32.69 (52.454) | 16.08 (54.920) | -18.75 (63.438) | -75.14 (84.820)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -12.25 (53.177) | -2.69 (76.234) | 18.23 (84.810) | -5.08 (77.809) | -54.79 (59.832)

35. Secondary Outcome: Change From Baseline In Large Low Density Lipoprotein Cholesterol (LDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Baseline, Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nmol/L
  Baseline | 367.42 (251.928) | 424.71 (336.502) | 578.57 (346.792) | 459.00 (341.699) | 639.36 (378.728)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | 16.42 (238.022) | -135.36 (140.673) | -138.69 (108.767) | -163.85 (183.861) | -219.64 (173.835)
  Change at Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 15 | -71.67 (265.452) | -198.31 (154.965) | -173.08 (158.586) | -248.25 (218.091) | -297.36 (201.235)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -26.50 (137.911) | -162.69 (170.876) | -237.00 (173.930) | -271.58 (219.097) | -311.36 (215.078)
  Change at Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 36 | -38.17 (164.092) | -93.15 (170.770) | -236.23 (180.758) | -244.75 (219.917) | -333.64 (266.184)
  Change at Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 50 | 18.83 (159.906) | -70.38 (111.722) | -177.46 (177.244) | -226.75 (161.785) | -337.00 (215.720)
  Change at Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 64 | -45.08 (227.314) | -114.31 (208.922) | -79.69 (168.660) | -147.75 (155.138) | -341.57 (243.742)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -50.08 (133.655) | -31.23 (254.307) | -108.15 (159.176) | -85.25 (91.821) | -215.43 (230.488)

36. Secondary Outcome: Change From Baseline In Total Low Density Lipoprotein Cholesterol (LDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Baseline, Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nmol/L
  Baseline | 1898.83 (393.934) | 1789.29 (297.035) | 1626.14 (474.106) | 1694.15 (439.012) | 1549.71 (332.241)
  Change at Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Change at Day 8 | -100.42 (326.272) | -598.00 (253.302) | -460.08 (351.468) | -664.00 (332.371) | -557.86 (245.049)
  Change at Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 15 | -87.67 (269.313) | -756.46 (300.314) | -658.08 (400.172) | -851.67 (447.423) | -790.14 (269.961)
  Change at Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 22 | -89.17 (344.100) | -877.62 (276.218) | -735.92 (462.348) | -1015.00 (482.252) | -846.71 (303.019)
  Change at Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 36 | -113.58 (299.598) | -345.46 (272.208) | -805.46 (413.417) | -986.75 (466.474) | -894.21 (284.814)
  Change at Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 50 | 63.00 (303.420) | -45.23 (128.264) | -278.23 (268.441) | -705.00 (486.227) | -879.50 (322.993)
  Change at Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 64 | -0.33 (287.226) | 10.62 (191.872) | -14.77 (231.884) | -309.25 (396.535) | -801.36 (354.429)
  Change at Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Change at Day 78 | -60.83 (285.233) | -105.62 (319.186) | -72.69 (364.420) | -143.42 (432.459) | -529.57 (294.496)

37. Secondary Outcome: Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Levels at Baseline, Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Baseline, Day 8, 15, 22, 36, 50, 64 and 78
Population: Pharmacodynamic analysis population was defined as all enrolled participants who received at least 1 dose of study medication and had atleast 1 pharmacodynamic parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
ng/mL
  Baseline | 48.83 (22.741) | 43.96 (23.731) | 43.07 (23.580) | 34.10 (20.316) | 44.12 (24.425)
  Day 8 | 48.53 (21.549) | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ).
  Day 15 | 50.42 (22.170) | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ).
  Day 22 | 52.58 (29.516) | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ).
  Day 36 | 51.80 (24.231) | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ).
  Day 50 | 48.21 (19.973) | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ).
  Day 64 | 51.95 (25.584) | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ).
  Day 78 | 43.75 (23.686) | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ). | NA (NA) — Data could not be evaluated since the value was below Lower Limit of Quantification (LLQ).

38. Secondary Outcome: C-Reactive Protein Levels at Day 8, 15, 21, 36, 57 and 78
Time Frame: Day 8, 15, 21, 36, 57 and 78
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
mg/dL
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 0.23 (0.252) | 0.26 (0.204) | 0.18 (0.251) | 0.42 (0.506) | 0.16 (0.191)
  Day 15: number analyzed (Participants) | 12 | 14 | 13 | 12 | 14
  Day 15 | 0.30 (0.385) | 0.23 (0.206) | 0.25 (0.433) | 0.38 (0.553) | 0.20 (0.293)
  Day 21: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 21 | 0.27 (0.320) | 0.23 (0.194) | 0.23 (0.441) | 0.32 (0.464) | 0.21 (0.364)
  Day 36: number analyzed (Participants) | 11 | 13 | 12 | 12 | 13
  Day 36 | 0.34 (0.407) | 0.27 (0.255) | 0.27 (0.450) | 0.28 (0.306) | 0.26 (0.541)
  Day 57: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 57 | 0.21 (0.205) | 0.36 (0.502) | 0.21 (0.368) | 0.51 (0.985) | 0.18 (0.220)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 0.32 (0.400) | 0.33 (0.522) | 0.21 (0.291) | 0.54 (1.175) | 0.15 (0.141)

39. Secondary Outcome: Small High Density Lipoprotein-Cholesterol (HDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: micromole/liter (umol/L)
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
micromole/liter (umol/L)
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 23.26 (3.147) | 22.79 (3.210) | 20.64 (7.390) | 19.74 (5.807) | 21.49 (5.767)
  Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 15 | 23.13 (5.511) | 24.04 (3.831) | 22.39 (6.412) | 19.04 (5.768) | 21.87 (7.229)
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 22.74 (5.162) | 23.67 (4.626) | 21.60 (6.865) | 21.57 (6.763) | 21.02 (6.531)
  Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 36 | 23.16 (5.582) | 23.33 (5.223) | 21.72 (5.804) | 19.18 (6.676) | 22.59 (5.060)
  Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 50 | 23.25 (3.395) | 23.73 (4.924) | 23.37 (5.005) | 22.83 (6.103) | 22.61 (8.649)
  Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 64 | 25.13 (4.747) | 23.02 (6.617) | 22.89 (5.298) | 20.73 (5.579) | 22.92 (7.777)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 22.79 (4.176) | 22.25 (6.245) | 21.85 (5.610) | 20.16 (5.633) | 21.11 (6.976)

40. Secondary Outcome: Medium High Density Lipoprotein-Cholesterol (HDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
umol/L
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 1.90 (2.158) | 4.24 (3.086) | 5.12 (3.778) | 6.24 (4.067) | 5.29 (5.057)
  Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 15 | 2.80 (2.888) | 4.88 (2.467) | 4.82 (3.408) | 8.69 (5.054) | 5.84 (6.642)
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 3.26 (2.394) | 5.60 (3.836) | 6.81 (5.102) | 5.71 (3.563) | 7.08 (6.606)
  Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 36 | 4.29 (3.516) | 4.75 (3.583) | 5.31 (3.738) | 8.34 (6.035) | 6.06 (4.500)
  Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 50 | 3.68 (3.615) | 3.48 (2.869) | 3.28 (3.059) | 4.94 (3.596) | 7.50 (7.664)
  Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 64 | 3.50 (3.254) | 2.82 (2.722) | 3.74 (3.358) | 4.73 (3.772) | 7.04 (6.034)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 3.65 (3.592) | 3.28 (3.006) | 2.88 (3.098) | 4.19 (4.274) | 5.37 (6.117)

41. Secondary Outcome: Large High Density Lipoprotein-Cholesterol (HDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
umol/L
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 5.88 (3.636) | 6.81 (3.963) | 7.97 (3.491) | 6.87 (4.608) | 8.08 (4.144)
  Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 15 | 5.90 (3.514) | 6.11 (3.684) | 9.05 (3.604) | 7.03 (3.833) | 8.36 (3.815)
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 6.23 (3.497) | 6.85 (3.152) | 7.93 (3.943) | 6.75 (3.544) | 8.88 (4.919)
  Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 36 | 5.70 (2.763) | 6.97 (4.091) | 8.25 (4.123) | 7.74 (4.124) | 8.94 (3.656)
  Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 50 | 5.95 (3.293) | 5.98 (3.452) | 7.58 (4.065) | 7.90 (4.608) | 9.06 (4.073)
  Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 64 | 5.78 (3.155) | 5.98 (2.471) | 7.47 (3.564) | 7.41 (5.359) | 7.65 (2.848)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 5.17 (2.934) | 5.61 (2.271) | 7.74 (3.788) | 7.16 (4.958) | 8.56 (3.747)

42. Secondary Outcome: Total High Density Lipoprotein-Cholesterol (HDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
umol/L
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 31.07 (5.339) | 33.84 (4.326) | 33.72 (5.344) | 32.85 (7.554) | 34.83 (5.854)
  Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 15 | 31.83 (6.791) | 35.03 (5.080) | 36.27 (5.541) | 34.77 (7.503) | 36.09 (7.021)
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 32.20 (5.874) | 36.13 (4.392) | 36.32 (5.852) | 34.02 (6.845) | 36.97 (5.193)
  Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 36 | 33.13 (6.369) | 35.04 (4.876) | 35.27 (4.077) | 35.28 (7.642) | 37.59 (4.453)
  Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 50 | 32.88 (4.380) | 33.21 (3.305) | 34.22 (4.704) | 35.69 (6.808) | 39.16 (5.797)
  Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 64 | 34.41 (6.210) | 31.84 (4.979) | 34.08 (3.930) | 32.88 (5.865) | 37.59 (4.620)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 31.61 (4.440) | 31.14 (5.035) | 32.48 (4.043) | 31.51 (6.288) | 35.01 (2.773)

43. Secondary Outcome: Small Very Low Density Lipoprotein-Cholesterol (VLDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nmol/L
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 48.02 (19.760) | 38.97 (17.319) | 36.84 (16.561) | 36.69 (18.980) | 28.94 (18.740)
  Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 15 | 54.04 (18.566) | 30.55 (13.832) | 29.98 (22.143) | 26.65 (12.759) | 23.56 (12.336)
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 50.14 (17.239) | 28.86 (11.540) | 20.91 (14.011) | 23.23 (10.315) | 20.94 (14.117)
  Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 36 | 55.32 (16.242) | 44.25 (18.962) | 24.22 (15.588) | 25.43 (14.978) | 21.39 (12.817)
  Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 50 | 50.04 (19.344) | 57.12 (20.032) | 34.65 (14.144) | 28.56 (16.992) | 24.69 (14.503)
  Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 64 | 51.82 (22.057) | 57.12 (22.475) | 42.09 (12.780) | 35.91 (16.296) | 18.81 (12.118)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 50.44 (24.319) | 48.44 (15.108) | 46.30 (90.153) | 39.72 (18.003) | 27.71 (17.448)

44. Secondary Outcome: Medium Very Low Density Lipoprotein-Cholesterol (VLDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nmol/L
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 43.84 (31.720) | 31.89 (16.142) | 21.82 (12.659) | 32.02 (20.966) | 34.56 (28.586)
  Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 15 | 45.18 (33.883) | 29.93 (12.067) | 31.38 (25.580) | 34.84 (26.305) | 33.91 (26.636)
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 42.08 (30.055) | 32.32 (16.184) | 35.10 (20.188) | 39.47 (22.121) | 30.62 (17.768)
  Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 36 | 54.42 (43.631) | 38.26 (25.474) | 19.35 (9.353) | 29.31 (18.029) | 26.48 (18.798)
  Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 50 | 40.91 (29.614) | 39.62 (26.490) | 25.31 (19.813) | 34.01 (20.440) | 25.04 (19.770)
  Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 64 | 46.29 (48.067) | 35.02 (23.457) | 21.05 (16.456) | 38.27 (28.436) | 24.48 (15.117)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 31.68 (26.579) | 33.54 (19.946) | 30.74 (24.781) | 38.25 (33.529) | 30.55 (35.729)

45. Secondary Outcome: Large Very Low Density Lipoprotein-Cholesterol (VLDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nmol/L
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 4.66 (7.571) | 3.91 (3.291) | 2.43 (3.119) | 5.18 (5.910) | 4.63 (8.128)
  Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 15 | 2.84 (3.086) | 3.69 (3.202) | 2.36 (2.425) | 5.58 (6.071) | 3.19 (4.364)
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 4.07 (4.367) | 3.65 (3.692) | 2.52 (3.384) | 2.75 (2.821) | 4.01 (7.348)
  Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 36 | 6.72 (7.795) | 3.85 (3.261) | 2.17 (2.615) | 4.27 (3.359) | 3.91 (6.648)
  Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 50 | 5.93 (6.572) | 3.25 (2.712) | 2.47 (3.347) | 5.57 (7.217) | 3.31 (4.728)
  Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 64 | 8.41 (12.714) | 3.42 (3.224) | 2.13 (3.096) | 6.33 (8.829) | 2.51 (3.305)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 9.00 (15.067) | 4.08 (3.494) | 2.34 (2.993) | 6.68 (9.279) | 2.89 (3.806)

46. Secondary Outcome: Total Very Low Density Lipoprotein-Cholesterol (VLDL-C) Particle Levels at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nmol/L
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 96.56 (37.874) | 74.79 (27.473) | 61.11 (26.738) | 73.92 (40.221) | 68.14 (37.104)
  Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 15 | 102.08 (40.769) | 64.16 (24.573) | 63.68 (44.340) | 67.07 (36.861) | 60.66 (33.367)
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 96.27 (42.925) | 64.85 (23.841) | 58.53 (26.727) | 65.47 (29.936) | 55.53 (23.928)
  Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 36 | 116.48 (59.693) | 86.36 (40.242) | 45.72 (20.487) | 58.99 (29.746) | 51.76 (26.621)
  Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 50 | 96.89 (39.372) | 100.00 (44.554) | 62.46 (29.705) | 68.13 (29.699) | 53.04 (31.259)
  Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 64 | 106.51 (66.108) | 95.55 (40.252) | 65.25 (27.024) | 80.51 (45.939) | 45.81 (24.781)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 91.11 (38.064) | 86.06 (31.763) | 79.37 (39.806) | 84.64 (50.216) | 61.16 (42.496)

47. Secondary Outcome: High Density Lipoprotein-Cholesterol (HDL-C) Particle Size at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nm
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 8.73 (0.454) | 8.81 (0.359) | 9.02 (0.421) | 8.88 (0.513) | 9.01 (0.427)
  Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 15 | 8.72 (0.356) | 8.75 (0.364) | 9.06 (0.371) | 8.95 (0.427) | 9.04 (0.425)
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 8.73 (0.379) | 8.84 (0.331) | 8.99 (0.362) | 8.92 (0.471) | 9.07 (0.412)
  Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 36 | 8.75 (0.406) | 8.85 (0.369) | 9.05 (0.470) | 9.03 (0.479) | 9.09 (0.342)
  Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 50 | 8.73 (0.398) | 8.77 (0.384) | 8.98 (0.419) | 8.95 (0.547) | 9.04 (0.403)
  Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 64 | 8.75 (0.303) | 8.77 (0.307) | 9.01 (0.441) | 8.96 (0.571) | 8.96 (0.386)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 8.68 (0.339) | 8.76 (0.263) | 9.05 (0.484) | 8.99 (0.507) | 9.08 (0.395)

48. Secondary Outcome: Very Low Density Lipoprotein-Cholesterol (VLDL-C) Particle Size at Day 8, 15, 22, 36, 50, 64 and 78
Time Frame: Day 8, 15, 22, 36, 50, 64 and 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 1.50 mg/kg
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 14
nm
  Day 8: number analyzed (Participants) | 12 | 14 | 13 | 13 | 14
  Day 8 | 48.57 (6.907) | 51.21 (5.290) | 50.15 (8.341) | 51.37 (6.934) | 50.07 (6.934)
  Day 15: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 15 | 48.13 (4.918) | 52.85 (5.284) | 53.57 (10.417) | 53.47 (8.371) | 50.54 (5.837)
  Day 22: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 22 | 52.42 (6.876) | 54.09 (6.152) | 54.28 (9.695) | 50.22 (4.799) | 53.95 (8.878)
  Day 36: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 36 | 51.42 (7.249) | 51.81 (6.030) | 53.69 (10.745) | 55.33 (9.556) | 52.40 (9.080)
  Day 50: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 50 | 51.57 (9.261) | 47.62 (4.463) | 53.62 (15.032) | 52.48 (9.738) | 54.14 (10.801)
  Day 64: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 64 | 50.51 (9.062) | 46.58 (6.099) | 48.60 (7.661) | 52.95 (8.965) | 51.74 (5.163)
  Day 78: number analyzed (Participants) | 12 | 13 | 13 | 12 | 14
  Day 78 | 52.17 (11.873) | 48.95 (4.820) | 49.41 (7.249) | 50.99 (8.967) | 49.63 (6.762)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Groups:
- PF-04950615 1.00 mg/kg: Participants recieved a single dose of PF-04950615 1.0 milligram/kilogram (mg/kg), intravenous (IV) infusion once on Day 1,8,15 and 22.
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 0.50 mg/kg | PF-04950615 1.00 mg/kg | PF-04950615 1.50 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/14 | 0/14 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 9/12 | 8/14 | 5/14 | 7/13 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | PF-04950615 0.25 mg/kg (N=14) | PF-04950615 0.50 mg/kg (N=14) | PF-04950615 1.00 mg/kg (N=13) | PF-04950615 1.50 mg/kg (N=14)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | PF-04950615 0.25 mg/kg (N=14) | PF-04950615 0.50 mg/kg (N=14) | PF-04950615 1.00 mg/kg (N=13) | PF-04950615 1.50 mg/kg (N=14)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Application site dermatitis (General disorders) | 0 | 1 | 0 | 0 | 0
Energy increased (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Puncture site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 2 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
QRS axis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 4 | 1 | 5
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.